CLINICAL TRIAL: NCT02335242
Title: Phase 2 Study of Sildenafil for the Treatment of Lymphatic Malformations
Brief Title: Sildenafil for the Treatment of Lymphatic Malformations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 23400; R01FD004372 (FDA)
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-10

CONDITIONS: Lymphatic Malformations; Lymphatic Diseases
Keywords: Sildenafil; Magnetic Resonance Imaging; Dermatology; Pediatrics
MeSH Terms: conditions — Lymphatic Abnormalities; Lymphatic Diseases | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo tablets (resembling Revatio) (Placebo Comparator): Placebo Drug: Placebo tablets (resembling Revatio)
  Interventions: Other: Placebo tablets (resembling Revatio)
- Sildenafil 20 mg tablets (Revatio) (Experimental): Active Drug: Sildenafil tablets (Revatio)
  Interventions: Drug: Sildenafil 20 mg tablets

INTERVENTIONS:
Drug: Sildenafil 20 mg tablets
  Arms: Sildenafil 20 mg tablets (Revatio)
Other: Placebo tablets (resembling Revatio)
  Arms: Placebo tablets (resembling Revatio)

SUMMARY:
A Phase 2 study to evaluate safety and efficacy of sildenafil taken orally to improve or resolve lymphatic malformations in children. Subjects may receive either placebo or treatment in an oral dosage with an open label extension for subjects who received placebo. The study treatment assignment will be randomized in a double blind fashion. MRI examination will evaluate change in lesion volume due to treatment. Other safety and efficacy measures will be taken through the 32-week study duration.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Lymphatic malformations (LMs) are localized areas of abnormal development of the lymphatic system that commonly occur in the head and neck of children. LMs are considered a rare or orphan disease which causes complications including pain, ulceration, secondary infection, infiltration of other organs, and death. Current therapies involve surgical excision or methods of chemical or physical destruction of portions of lesions. No therapies are uniformly effective and all have the risk of significant adverse events. We recently witnessed almost complete resolution of a LM lesion in a child who was treated with sildenafil oral therapy for pulmonary arterial hypertension. We have subsequently evaluated additional subjects who improved with sildenafil. The goal of this clinical research trial is to document the benefit or absence of benefit of sildenafil therapy for LMs and identify which type of patient will benefit from sildenafil. This study is a double-blind placebo-controlled trial which involves precise documentation of volume changes associated with therapy or placebo by using MRI segmentation techniques. We will also observe and document the clinical response to sildenafil or placebo using clinical evaluation scores and surveys. The results of the study should identify characteristics of LM lesions which may suggest a beneficial response to sildenafil therapy. Sildenafil has very low risk of side effects in the dosage used in this trial. Documentation of an effective response of LMs to sildenafil will accelerate the interest in, and the ability to understand, the mechanisms of LM formation and treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* Be legally authorized representative of subjects willing and able to give consent. Assent obtained for subjects 7 - 10 years old.
* Be between the ages of 6 months - 10 years of age at the time of entry into the study.
* Be at the minimum weight of 8 kg at the time of enrollment.
* Be required to have the clinical diagnosis of lymphatic malformation that appears to be over 3 cm in greatest diameter in order to be evaluated for entry. A review of a previous MRI examination may help confirm the entry criteria on subjects selected to come to Stanford for the MRI screening.
* Have the lymphatic malformation cause enough disability for the subject that requires them to consider systemic therapy.
* For female subjects: must not be pregnant or breast-feeding.
* Have a parent or legally authorized representative willing and able to ensure subject is present for all required study visits.
* Have a required MRI examination to confirm that the lymphatic malformation is present and is greater than 3 cm in diameter in order for the subjects to receive medication, which happens during the initial screening evaluation portion of the trial.
* Have no contraindications for the use of sildenafil.
* Have a normal eye examination.
* Have normal liver and kidney function.
* Have no contraindication to MRI examinations such as metal implants, etc.
* Not be a smoker.

Exclusion Criteria:

A Subject with any of the following criteria is not eligible for inclusion in this study:

* Medically unstable health status that may interfere with his/her ability to complete the study.
* Has one or more of the following medical conditions:

Hepatic impairment, severe renal impairment, lymphedema conditions such as Milroy disease, Meige lymphedema, Hennekam syndrome, Njolstad syndrome, Aagenaes syndrome, and Fabry disease, hypotension or at risk for hypotension, seizures or history of seizures, any significant cardiovascular risk factors and any condition which requires participants to use nitric oxide donors or nitrates in any form, underlying anatomic or vascular risk factor for developing non-arteritic anterior ischemic optic neuropathy (NAION) including low ocular cup to disc ratio, diabetes, hypertension, coronary artery disease, or hyperlipidemia Participants with Down syndrome, Turner syndrome and Noonan syndrome will be considered on a case-by-case basis.

* Has received at least one of the following medications contraindicated in association with sildenafil within 15 days of inclusion:

  * Organic nitrates in any form, either regularly or intermittently -- Consistent with its known effects on the nitric oxide/cGMP pathway, sildenafil was shown to potentiate the hypotensive effects of nitrates.
  * Ritonavir and other Potent CYP3A Inhibitors --- Concomitant use of REVATIO with ritonavir and other potent CYP3A inhibitors is not recommended.
  * Alpha-blockers --- co-administering alpha-blockers with REVATIO because of additive blood pressure-lowering effects
  * Amlodipine
  * Cimetidine
* Requires concomitant use of potent cytochrome P450 3A4 inhibitors (such as ketoconazole, itraconazole, erythromycin, saquinavir), or concomitant use of ritonavir. Also excluded are concomitant use of organic nitrates, alpha-blockers, amlodipine, or cimetidine.
* Cannot confirm that the lesion is a lymphatic malformation or the lymphatic malformation is less than 3 cm in its greatest diameter during the MRI screening.
* Has had extensive prior surgery or sclerotherapy to treat LM such that scarring may interfere with evaluation and treatment effect of sildenafil.
* Have had recurrent infection and significant scarring of the lesion secondary to infection to such an extent that the that scarring may interfere with evaluation and treatment effect of sildenafil
* Known to have an allergy to sildenafil.
* Has ulcerated or currently infected LMs.
* Has diagnosis of the soft tissue tumor as LM not clinically certain.
* Participating in another clinical study which may interfere.
* Has a history of priapism or is diagnosed with sickle cell anemia or any other disorder which may predispose to priapism.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-05-23 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Teng, MD, PhD, Principal Investigator — Stanford School of Medicine
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - University of Colorado, Denver, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No
The IPD will only be shared de-identified to our study staff and human subjects approved subsites. These results will eventually be published, but will be completed around 2022.

REFERENCES:
- [Background] Abrams D, Schulze-Neick I, Magee AG. Sildenafil as a selective pulmonary vasodilator in childhood primary pulmonary hypertension. Heart. 2000 Aug;84(2):E4. doi: 10.1136/heart.84.2.e4. PMID 10908271
- [Background] Barst RJ, Ivy DD, Gaitan G, Szatmari A, Rudzinski A, Garcia AE, Sastry BK, Pulido T, Layton GR, Serdarevic-Pehar M, Wessel DL. A randomized, double-blind, placebo-controlled, dose-ranging study of oral sildenafil citrate in treatment-naive children with pulmonary arterial hypertension. Circulation. 2012 Jan 17;125(2):324-34. doi: 10.1161/CIRCULATIONAHA.110.016667. Epub 2011 Nov 29. PMID 22128226
- [Background] Berk DR, Berk EJ, Bruckner AL. A novel method for calculating the volume of hemangiomas. Pediatr Dermatol. 2011 Jul-Aug;28(4):478-82. doi: 10.1111/j.1525-1470.2011.01498.x. PMID 21793894
- [Background] Blei F. Congenital lymphatic malformations. Ann N Y Acad Sci. 2008;1131:185-94. doi: 10.1196/annals.1413.016. PMID 18519970
- [Background] Churchill P, Otal D, Pemberton J, Ali A, Flageole H, Walton JM. Sclerotherapy for lymphatic malformations in children: a scoping review. J Pediatr Surg. 2011 May;46(5):912-22. doi: 10.1016/j.jpedsurg.2011.02.027. PMID 21616252
- [Background] de Graaf M, Breur JMPJ, Raphael MF, Vos M, Breugem CC, Pasmans SGMA. Adverse effects of propranolol when used in the treatment of hemangiomas: a case series of 28 infants. J Am Acad Dermatol. 2011 Aug;65(2):320-327. doi: 10.1016/j.jaad.2010.06.048. Epub 2011 May 20. PMID 21601311
- [Background] Fisher R, Partington A, Dykes E. Cystic hygroma: comparison between prenatal and postnatal diagnosis. J Pediatr Surg. 1996 Apr;31(4):473-6. doi: 10.1016/s0022-3468(96)90477-7. PMID 8801294
- [Background] Frieden IJ, Drolet BA. Propranolol for infantile hemangiomas: promise, peril, pathogenesis. Pediatr Dermatol. 2009 Sep-Oct;26(5):642-4. doi: 10.1111/j.1525-1470.2009.00977.x. No abstract available. PMID 19840341
- [Background] Fuchsmann C, Quintal MC, Giguere C, Ayari-Khalfallah S, Guibaud L, Powell J, McCone C, Froehlich P. Propranolol as first-line treatment of head and neck hemangiomas. Arch Otolaryngol Head Neck Surg. 2011 May;137(5):471-8. doi: 10.1001/archoto.2011.55. PMID 21576558
- [Background] Gallagher PG, Mahoney MJ, Gosche JR. Cystic hygroma in the fetus and newborn. Semin Perinatol. 1999 Aug;23(4):341-56. doi: 10.1016/s0146-0005(99)80042-1. PMID 10475547
- [Background] Greene AK, Perlyn CA, Alomari AI. Management of lymphatic malformations. Clin Plast Surg. 2011 Jan;38(1):75-82. doi: 10.1016/j.cps.2010.08.006. PMID 21095473
- [Background] Howarth ES, Draper ES, Budd JL, Konje JC, Clarke M, Kurinczuk JJ. Population-based study of the outcome following the prenatal diagnosis of cystic hygroma. Prenat Diagn. 2005 Apr;25(4):286-91. doi: 10.1002/pd.1100. PMID 15849783
- [Background] Karatza AA, Bush A, Magee AG. Safety and efficacy of Sildenafil therapy in children with pulmonary hypertension. Int J Cardiol. 2005 Apr 20;100(2):267-73. doi: 10.1016/j.ijcard.2004.09.002. PMID 15823634
- [Background] Leaute-Labreze C, Dumas de la Roque E, Hubiche T, Boralevi F, Thambo JB, Taieb A. Propranolol for severe hemangiomas of infancy. N Engl J Med. 2008 Jun 12;358(24):2649-51. doi: 10.1056/NEJMc0708819. No abstract available. PMID 18550886
- [Background] Pfizer. (2007).
- [Background] Redondo P, Aguado L, Martinez-Cuesta A. Diagnosis and management of extensive vascular malformations of the lower limb: part I. Clinical diagnosis. J Am Acad Dermatol. 2011 Nov;65(5):893-906; quiz 907-8. doi: 10.1016/j.jaad.2010.12.047. PMID 22000870
- [Background] Sans V, de la Roque ED, Berge J, Grenier N, Boralevi F, Mazereeuw-Hautier J, Lipsker D, Dupuis E, Ezzedine K, Vergnes P, Taieb A, Leaute-Labreze C. Propranolol for severe infantile hemangiomas: follow-up report. Pediatrics. 2009 Sep;124(3):e423-31. doi: 10.1542/peds.2008-3458. Epub 2009 Aug 10. PMID 19706583
- [Background] Shekerdemian LS, Ravn HB, Penny DJ. Intravenous sildenafil lowers pulmonary vascular resistance in a model of neonatal pulmonary hypertension. Am J Respir Crit Care Med. 2002 Apr 15;165(8):1098-102. doi: 10.1164/ajrccm.165.8.2107097. PMID 11956051
- [Background] Wang P, Wu P, Egan RW, Billah MM. Identification and characterization of a new human type 9 cGMP-specific phosphodiesterase splice variant (PDE9A5). Differential tissue distribution and subcellular localization of PDE9A variants. Gene. 2003 Sep 18;314:15-27. doi: 10.1016/s0378-1119(03)00733-9. PMID 14527714
- [Background] Whimster IW. The pathology of lymphangioma circumscriptum. Br J Dermatol. 1976 May;94(5):473-86. doi: 10.1111/j.1365-2133.1976.tb05134.x. PMID 1268059

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 78 individuals were assessed for eligibility; 22 were enrolled, and 19 were randomized to a study arm.
Groups:
- Double-Blind Placebo Then Open-Label Sildenafil: Placebo (resembling Revatio) for 20 weeks. Participants randomized to placebo had the option to enter a 20-week open-label phase to receive active sildenafil (Revatio) for 20 weeks three times daily (weight-based: 10 mg TID for participants weighing 8-20 kg; 20 mg TID for participants weighing >20 kg), followed by a 12 week follow-up period.
- Double-Blind Sildenafil: Sildenafil (Revatio) for 20 weeks three times daily (weight-based: 10 mg TID for participants weighing 8-20 kg; 20 mg TID for participants weighing >20 kg), followed by a 12-week follow-up period.
Period: Randomized Phase (20 Weeks)
Arm/Group | Double-Blind Placebo Then Open-Label Sildenafil | Double-Blind Sildenafil
Started | 8 | 11
Completed | 7 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Open-label Phase (20 Weeks)
Arm/Group | Double-Blind Placebo Then Open-Label Sildenafil | Double-Blind Sildenafil
Started | 6 (1 participant did not continue to the open-label phase.) | 0 (Participants in the sildenafil group did not enter the open-label phase, but proceeded to the follow-up period.)
Completed | 6 | 0
Not Completed | 0 | 0
Period: Follow-up Period (12 Weeks)
Arm/Group | Double-Blind Placebo Then Open-Label Sildenafil | Double-Blind Sildenafil
Started | 6 | 11
Completed | 4 | 10
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Discontinued intervention | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Placebo Then Open-Label Sildenafil | Double-Blind Sildenafil | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 11 | 19
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data are available for only 6 participants in the placebo group.
  Participants
    number analyzed (Participants) | 6 | 11 | 17
    Hispanic or Latino | 1 | 5 | 6
    Not Hispanic or Latino | 5 | 6 | 11
    Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race data are available for only 6 participants in the placebo group.
  Participants
    African American: number analyzed (Participants) | 6 | 11 | 17
    African American | 1 | 0 | 1
    Asian: number analyzed (Participants) | 6 | 11 | 17
    Asian | 0 | 2 | 2
    Indian: number analyzed (Participants) | 6 | 11 | 17
    Indian | 1 | 0 | 1
    White: number analyzed (Participants) | 6 | 11 | 17
    White | 2 | 3 | 5
    More than one race: number analyzed (Participants) | 6 | 11 | 17
    More than one race | 1 | 1 | 2
    Unknown/Not reported: number analyzed (Participants) | 6 | 11 | 17
    Unknown/Not reported | 1 | 5 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 11 | 19
Lesion volume [Median (Full Range); unit: mm^3] — Population: Baseline lesion volume data are available for only 6 participants in the placebo group.
  mm^3
    number analyzed (Participants) | 6 | 11 | 17
    (all) | 49 [10 to 280] | 144 [49 to 856] | 87 [10 to 856]

OUTCOME MEASURES:

1. Primary Outcome: Change in Lesion Volume of the Test Medication as Evaluated by MRI Examination.
Description: Participants will be followed for the duration of the study, an expected average of 20 weeks.
Time Frame: Baseline, week 20
Population: Participants who completed each treatment period are included in the analysis
Measure: Mean (Standard Deviation); unit: percentage of volume
Groups:
- Double-Blind Placebo: Placebo (resembling Revatio) for 20 weeks, followed by a 12 week follow-up period.
- Open-Label Sildenafil: Participants who complete placebo then receive active sildenafil (Revatio) for 20 weeks three times daily (weight-based: 10 mg TID for participants weighing 8-20 kg; 20 mg TID for participants weighing >20 kg), followed by a 12 week follow-up period.
Arm/Group | Double-Blind Placebo | Open-Label Sildenafil | Double-blind Sildenafil
Number analyzed (Participants) | 7 | 6 | 10
percentage of volume | 5.89 (13.5) | -8.54 (12.1) | -0.642 (18.3)

2. Secondary Outcome: Change in Subject's Assessment of Change in Lymphatic Malformation Overall Score
Description: Subject's evaluation of the overall change in lymphatic malformation. Participants will be followed from baseline to 20 weeks.
  Patients rated change as no improvement, minimal improvement (1-25% change), fair improvement (25-50% change), good improvement (50-75% change), and excellent improvement (75-100% change).
Time Frame: Baseline, week 20
Population: Participants with data at both baseline and week 20 are included in the analysis
Measure: Count of Participants; unit: Participants
Groups:
- Double-Blind Placebo: Placebo (resembling Revatio) for 20 weeks.
- Double-Blind Sildenafil: Sildenafil (Revatio) for 20 weeks three times daily (weight-based: 10 mg TID for participants weighing 8-20 kg; 20 mg TID for participants weighing >20 kg).
Arm/Group | Double-Blind Placebo | Double-Blind Sildenafil
Number analyzed (Participants) | 5 | 8
Participants
  No improvement | 1 | 2
  Minimal improvement | 2 | 4
  Fair improvement | 0 | 1
  Good improvement | 2 | 1
  Excellent improvement | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 52 weeks in the Placebo then Open-Label Sildenafil group, and up to 32 weeks in the Sildenafil group
Groups:
- Open-Label Sildenafil: Participants who complete placebo then receive active sildenafil (Revatio) for 20 weeks three times daily (weight-based: 10 mg TID for participants weighing 8-20 kg; 20 mg TID for participants weighing >20 kg).
Arm/Group | Double-Blind Placebo | Open-Label Sildenafil | Double-Blind Sildenafil
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 8/8 | 5/6 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Placebo (N=8) | Open-Label Sildenafil (N=6) | Double-Blind Sildenafil (N=10)
Cold (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Abdominal pain/bloating (Gastrointestinal disorders) | 0 | 1 | 2
Nausea/vomit (Gastrointestinal disorders) | 2 | 1 | 4
Loose stool/increase bowel movement (Gastrointestinal disorders) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Acute gastroenteritis/viral gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 1
Headaches (Nervous system disorders) | 0 | 2 | 5
Fever (General disorders) | 5 | 0 | 1
Intermittent flushing (Vascular disorders) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Only 1 of 4 planned sites participated in this trial; the study did not meet its planned enrollment and the results are underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT02335242/Prot_SAP_000.pdf